CLINICAL TRIAL: NCT07310199
Title: Pharmacist-Led Transition of Care Program in the Emergency Department (Pharm TOC-ED): A Pilot Randomized, Parallel-Group, Open-Label Trial With Embedded Process Evaluation
Brief Title: Pharmacist-Led Transition of Care Program in the Emergency Department (Pharm TOC-ED): A Pilot Trial
Acronym: PharmTOC-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Muhammad Abdul Hadi (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dr. Muhammad Abdul Hadi, Associate Professor of Clinical Pharmacy and Practice, Qatar University
Organization: Qatar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2394800-1; CG 838 (Other Grant/Funding Number: Qatar University)
Record Dates: First submitted 2025-12-14; First posted 2025-12-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transitional Care
Keywords: transition of care; Pharmacy services; Emergency Department
MeSH Terms: conditions — Emergencies | interventions — RHBDF2 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Usual Care) (No Intervention): Patients in this group will receive standard care in accordance with Hamad Medical Corporation's (HMC) policies and practices. Currently, case review by clinical pharmacists for all ED patients at the study site is not part of routine care. Medication review, reconciliation, discharge education, and follow-up are typically managed by ED-physicians and nurses. Clinical pharmacists may be consulted, depending on availability, for complex or selected cases only. Control group patients will not be denied pharmacist-led TOC services when deemed necessary as part of routine clinical judgment. These instances will be recorded, including the reason, nature, and timing of the care provided by the pharmacist.
- Multi-faceted pharmacist-led transition of care (ToC) program (Intervention) (Active Comparator): Participants receive usual care plus a pharmacist-led transition of care (ToC) program, which includes medication review, reconciliation, discharge counseling, coordination of follow-up, and post-discharge pharmacist visits.
  Interventions: Behavioral: Multi-faceted pharmacist-led transition of care (ToC) program

INTERVENTIONS:
Behavioral: Multi-faceted pharmacist-led transition of care (ToC) program — The pharmacist-led transition of care (ToC) intervention begins once a patient is deemed ready for ED discharge. ED pharmacists conduct a comprehensive discharge medication review, identify and resolve medication therapy problems, and document recommendations in the electronic health record (EHR). They perform discharge medication reconciliation, generate the best possible medication list, and correct any discrepancies. Pharmacists provide structured medication counseling using teach-back and address adherence barriers. Discharge planning includes scheduling post-discharge follow-up in a pharmacist-led medication therapy management clinic and delivering a standardized handover to ambulatory pharmacists. Patients receive two post-discharge follow-up visits within 7 and 14 days, during which pharmacists reassess medications, resolve new or ongoing issues, provide education, and coordinate additional care when needed. All activities follow standardized documentation procedures.
  Arms: Multi-faceted pharmacist-led transition of care (ToC) program (Intervention)

SUMMARY:
When patients leave the emergency department, mistakes with their medications are common and can lead to complications or hospital readmissions. Pharmacists are trained to help prevent these problems, but pharmacist-led transition of care services are not routinely provided in emergency departments.

This study is a small pilot randomized controlled trial designed to see whether a pharmacist-led transition of care program can be carried out successfully in the emergency department at Al-Wakra Hospital. The study will help determine if a larger trial is feasible in the future.

Patients who are being discharged home from the emergency department and meet the study criteria will be invited to participate. Those who agree will be randomly assigned to one of two groups:

Usual care, or Usual care plus the pharmacist-led transition of care program The pharmacist-led program includes reviewing the discharge prescription, checking and updating the medication list, providing medication education, arranging follow-up with a pharmacist-run clinic, communicating with outpatient pharmacists, and following up with the patient after discharge.

The pilot trial will help determine how many patients are eligible, how many agree to participate, how well the intervention can be delivered in the emergency department, and whether patients and staff find it acceptable. The results will be used to plan a larger study that will test whether this program can reduce healthcare use after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 years or more) discharged from the ED with at least one of the following:
* Polypharmacy: Five or more scheduled prescription medications for chronic illnesses (i.e., chronic maintenance medications, even if such medications were not refilled during the index ED visit)
* Discharged with a new prescription of high-risk medication, including:
* Drugs with the potential of withdrawal symptoms upon abrupt discontinuation such as antipsychotics, antiepileptics, antidepressants, and tapering glucocorticoids.
* Insulin (initiation or intensification of therapy)
* Oral hypoglycemic agents
* Visiting ED for an exacerbation of chronic illness (e.g., exacerbation of asthma, COPD, CHF, uncontrolled diabetes mellitus, hypertension urgency, uncontrolled epilepsy)

Exclusion Criteria:

* The following patients will be excluded:
* Presenting with acute minor illnesses
* Lack of decision-making capacity (including documented moderate or severe dementia, altered mental status, unstable psychiatric illness, altered consciousness level, lack of orientation to person/place/time as reported in EHR, delirium, patients seen in the ED for a psychiatric evaluation)
* Language barrier, i.e., inability to communicate in either English or Arabic as the intervention will be provided by English/Arabic speaking clinical pharmacists
* Expected length of stay in Qatar of <30 days post discharge (including transit passengers)
* Substance use disorders (e.g., alcoholism, opioid dependency) or drug-seeking behavior, as reported in EHR
* Prisoners who are serving an active sentence
* Patients presenting for non-medical, socially driven reasons (e.g., seeking shelter, support, or resources) with no identifiable acute medical condition, and known to the ED team as recurrent visitors.
* Discharge to a location other than home (e.g., patients transferred to another hospital, long-term or skilled nursing facility)
* Study pharmacists unavailable to deliver the intervention if the patients were randomized to the intervention arm
* Pregnant women
* Patients seen for trauma or planned surgery
* Terminally ill patients
* Patients discharged from ED with watchful waiting (e.g., expected to be readmitted for an intervention such as surgical intervention if conservative management failed)
* Patients who are admitted to the hospital after enrollment (i.e., following consent but prior to ED discharge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate among screened patients | At baseline (Day 1)
  Proportion of screened emergency department (ED) patients who meet all inclusion criteria and none of the exclusion criteria for the pilot trial.
Recruitment rate among eligible patients | At baseline (Day 1)
  Proportion of eligible patients who agree to participate, provide informed consent, and are randomized into the trial.
Retention rate at post-discharge follow-up | Intervention arm: Day 7, Day 14, and Day 30 after ED discharge, Control arm: Day 30 after ED discharge
  Proportion of enrolled patients who: (a) in the intervention group, attend pharmacist-led follow-up visits at 7 and 14 days after ED discharge; and (b) in both groups, complete the 30-day follow-up phone call.
Intervention fidelity: receipt of all ToC program components | Through day 30 after ED discharge
  Proportion of participants in the intervention arm who receive all prespecified components of the pharmacist-led transition of care intervention (discharge medication review, discharge medication reconciliation, patient counseling, discharge planning, and post-discharge follow-up).

SECONDARY OUTCOMES:
Proportion of patients with ≥1 unintentional medication discrepancy | Through day 30 after ED discharge
  Proportion of patients with at least one unintentional medication discrepancy identified by the clinical pharmacist at ED discharge and during post-discharge follow-up visits.
Number and types of unintentional medication discrepancies | Through Day 30 after ED discharge
  Total number, mean number per patient, and types of unintentional medication discrepancies identified by the clinical pharmacist at ED discharge and during post-discharge follow-up visits.
Proportion of patients with ≥1 medication therapy problem (MTP) | Through Day 30 after ED discharge
  Proportion of patients with at least one medication therapy problem identified by the clinical pharmacist at ED discharge and during post-discharge follow-up visits.
Number and types of medication therapy problems | Through Day 30 after ED discharge
  Total number, mean number per patient, and types of medication therapy problems identified by the clinical pharmacist at ED discharge and during post-discharge follow-up visits.
Resolution of medication discrepancies and medication therapy problems | Through Day 30 after ED discharge
  Proportion of identified medication discrepancies and medication therapy problems that are resolved before ED discharge, resolved during post-discharge follow-up, or remain unresolved at the end of follow-up.
Unplanned healthcare utilization within 30 days | Through Day 30 after ED discharge
  Proportion of patients with a composite outcome of unplanned ED revisit and/or unplanned hospital admission for any acute health problem within 30 days of discharge from the index ED visit. Elective admissions and scheduled outpatient visits are excluded.
ED revisit or hospital admission related to index ED presentation | Through Day 30 after ED discharge
  Proportion of patients with an ED revisit and/or hospital admission determined to be related to the index ED presentation within 30 days of discharge.
Medication-related ED visits or hospital admissions | Through Day 30 after ED discharge
  Proportion of patients with medication-related ED revisits and/or hospital admissions within 30 days of discharge, identified using AT-HARM10 screening followed by adjudication by a clinical pharmacist and physician.
Patient satisfaction with pharmacist-led ToC intervention | Day 30 after discharge
  Patient satisfaction with pharmacist-led transition of care interventions assessed using the Medication Management Patient Satisfaction Survey (MMPSS).

CONTACTS AND LOCATIONS:
Locations (1):
- Al- Wakra Hospital- Hamad Medical Corporation, Al Wakrah, Qatar

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team. Data will be analyzed and reported in aggregate form only, in accordance with institutional and ethical approvals.